CLINICAL TRIAL: NCT01204554
Title: Microcirculation in Perforator Flaps. Enhancing Tissue Survival
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Dr. Haris Mesic, Oslo University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08/223b.2008/3837 (REK)
Record Dates: First submitted 2010-09-06; First posted 2010-09-17 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Reconstructive Surgery; Microcirculation
Keywords: perforator flaps
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Indocyanine green (ICG) — a water-soluble dye that binds to plasma proteins and remains in the intravascular space after intravenous injection.ICG has a normal plasma half life of 3-4 min. Dosage planned is 0 .5 mg/kg dose of ICG resolved in 5 % dextrose 2 mg /ml.

SUMMARY:
The aim of the present study is to assess the microcirculatory changes in the distal part of the perforator flap using ICG fluorescence angiography.

DETAILED DESCRIPTION:
Perforator flaps are increasingly used in reconstructive surgery both as pedicled and free flaps, mostly because of reduced donor site morbidity and superior aesthetic result. However, the there is still much to learn about the hemodynamic changes within these flaps.The aim of the present study is to assess the microcirculatory changes in the distal part of the perforator flap using ICG fluorescence angiography.

ELIGIBILITY:
Inclusion Criteria:

* patients submitted to elective abdominoplasty

Exclusion Criteria:

* body mass index < 30 kg/m2
* morbidly obese
* patients with comorbidity such as diabetes
* vascular disease
* smokers
* patients < 18 years, and patients using anti-coagulant therapy
* pregnant
* severe hepatic insufficiency were excluded and a history of allergic reactions to ICG and iodide.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Mean pixel intensity using dynamic laser-induced-fluorescence-videoangiography | dec. 2008--des 2010
  Perfusion measurements were conducted intraoperatively by assessing microcirculation using the technique of dynamic laser-induced-fluorescence-videoangiography (IC-VIEW, PULSION Medical Systems AG, Munich, Germany).

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway